CLINICAL TRIAL: NCT01223469
Title: A Prospective Safety, Performance and Preliminary Effectiveness, Multi-centre, Clinical Investigation Using the Irrigated TactiCath™ Percutaneous Ablation Catheter for the Treatment of Supra-Ventricular Tachyarrhythmia Using RF Ablation
Brief Title: TOCCATA - Touch+™ for Catheter Ablation
Acronym: TOCCATA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Endosense (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VP-001 147
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Atrial Fibrillation; Tachycardia, Supraventricular
Keywords: Atrial Fibrillation; Supraventricular Tachycardia; Contact Force; RF Ablation; Radiofrequency; Pulmonary Vein Isolation; Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Tachycardia, Supraventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atrial Fibrillation (Experimental)
  Interventions: Device: Contact force assisted irrigated RF ablation
- Right-sided Supraventricular Tachycardia (Experimental)
  Interventions: Device: Contact force assisted irrigated RF ablation

INTERVENTIONS:
Device: Contact force assisted irrigated RF ablation — radiofrequency ablation of atrial fibrillation or SVT
  Other Names: TactiCath®; TactiSys®

SUMMARY:
The main objective of this study is to demonstrate the clinical safety of a contact force sensing RF ablation catheter when used for the treatment of supraventricular tachycardia and atrial fibrillation. In addition, the study will characterize the use and value of contact force measurement during ablation, and the long term success (12 months) of the ablation procedure using this technology.

DETAILED DESCRIPTION:
Safety: The primary safety endpoint assesses the incidence of procedure or device related SAEs from procedure to 7 (±1) days post-procedure or hospital discharge, whichever is longer, for patients with right-sided SVT or 3 months (±2 weeks) post-procedure for patients with atrial fibrillation. Secondary safety objectives were to demonstrate safety (operative and post-operative complications) over the 12 months post-procedure.

Performance: The primary performance endpoint is to demonstrate successful catheter deployment, irrigation and ablation at the target area during supra-ventricular cardiac ablation. The secondary performance endpoint is to demonstrate successful and effective contact force reading between catheter tip and heart wall during mapping and ablation at all locations and all angulations.

Efficacy: Secondary effectiveness objectives will consider acute and chronic elimination of the target arrhythmia, the cost-effectiveness of the system and procedure-related parameters

ELIGIBILITY:
Inclusion Criteria:

* Patients with right-sided SVT (including: atrioventricular nodal re entry tachycardia [AVNRT], accessory pathway Wolff Parkinson White [WPW] syndrome, atrial tachycardia or isthmus-dependent atrial flutter) or paroxysmal atrial fibrillation

Exclusion Criteria:

* Recent (within 3 months) cardiac events including myocardial infarction, acute coronary syndrome, percutaneous coronary intervention, or valve or coronary bypass graft surgery
* Moderate or severe structural heart disease (ventricular dysfunction or valve disease) as demonstrated by transthoracic (TTE) or transesophageal echocardiogram (TEE) of all four chambers of the heart
* Known cerebrovascular disease, including a history of stroke or transient ischemic attack
* Left ventricular ejection fraction of <35%
* Previous heart ablation procedure (surgical or catheter) to the target chamber

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2008-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Heinz Kuck, Prof, Principal Investigator — Asklepios Klinik St. Georg, Hamburg, Germany

REFERENCES:
- [Result] Reddy VY, Shah D, Kautzner J, Schmidt B, Saoudi N, Herrera C, Jais P, Hindricks G, Peichl P, Yulzari A, Lambert H, Neuzil P, Natale A, Kuck KH. The relationship between contact force and clinical outcome during radiofrequency catheter ablation of atrial fibrillation in the TOCCATA study. Heart Rhythm. 2012 Nov;9(11):1789-95. doi: 10.1016/j.hrthm.2012.07.016. Epub 2012 Jul 20. PMID 22820056
- [Result] Kuck KH, Reddy VY, Schmidt B, Natale A, Neuzil P, Saoudi N, Kautzner J, Herrera C, Hindricks G, Jais P, Nakagawa H, Lambert H, Shah DC. A novel radiofrequency ablation catheter using contact force sensing: Toccata study. Heart Rhythm. 2012 Jan;9(1):18-23. doi: 10.1016/j.hrthm.2011.08.021. Epub 2011 Aug 26. PMID 21872560
- See also: Reddy VY, et. al, The relationship between contact force and clinical outcome during radiofrequency catheter ablation of atrial fibrillation in the TOCCATA study.Heart Rhythm. 2012 Nov;9(11):1789-95 — http://www.ncbi.nlm.nih.gov/pubmed/22820056
- See also: Kuck KH, et.al; A novel radiofrequency ablation catheter using contact force sensing: Toccata study. Heart Rhythm. 2012 Jan;9(1):18-23 — http://www.ncbi.nlm.nih.gov/pubmed/21872560

RESULTS

PARTICIPANT FLOW:
Groups:
- Atrial Fibrillation: Contact force assisted irrigated RF ablation: radiofrequency ablation of atrial fibrillation.
- Right-sided Supraventricular Tachycardia: Contact force assisted irrigated RF ablation: radiofrequency ablation of SVT
Period: Overall Study
Arm/Group | Atrial Fibrillation | Right-sided Supraventricular Tachycardia
Started | 34 | 43
Completed | 34 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atrial Fibrillation | Right-sided Supraventricular Tachycardia | Total
Number analyzed (Participants) | 34 | 43 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 11 | 20
  >=65 years | 25 | 32 | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 23 | 29 | 52

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Operative and Post-operative Serious Adverse Events
Description: For Right SVT patients 7 days (±1 day) following the index procedure or until hospital discharge whichever is longer.
  For AF patients 3 months (±2 weeks)following the index procedure.
Time Frame: 3 months for AF arm; 7 days for the right SVT arm
Measure: Number; unit: participants
Arm/Group | Atrial Fibrillation | Right-sided Supraventricular Tachycardia
Number analyzed (Participants) | 34 | 43
participants | 4 | 1

ADVERSE EVENTS:
Arm/Group | Atrial Fibrillation | Right-sided Supraventricular Tachycardia
Serious Adverse Events (participants affected / at risk) | 4/34 | 1/43
Other Adverse Events (participants affected / at risk) | 0/34 | 0/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atrial Fibrillation (N=34) | Right-sided Supraventricular Tachycardia (N=43)
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) — In the SVT arm, the SAE was a sinus bradycardia, followed by pacemaker implantation in a patient treated for atrial flutter with the study device and with a standard ablation catheter for concomitant RA arrhythmias.
Tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Groin Bleeding (Vascular disorders) | 1 (1) | 0 (0)
Stroke (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No